CLINICAL TRIAL: NCT01816841
Title: The Role of Direct Visual Fluorescence in Oral Examination
Brief Title: Direct Visual Fluorescence in Finding Oral Cancer in High-Risk Patients and Patients Undergoing Routine Dental Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Kristin McNamara, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OSU-08095; NCI-2012-02017 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Lip and Oral Cavity Squamous Cell Carcinoma; Oral Cavity Verrucous Carcinoma; Stage 0 Lip and Oral Cavity Cancer; Tongue Cancer
Keywords: Direct Visual Fluorescense; Oral Examination; oral cancer
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia; Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms; Tongue Neoplasms | interventions — Optical Imaging; Biopsy; Restraint, Physical; Independent Medical Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diagnostic (COE and DVFE)- Arm I (Experimental): Arm I - Patients undergo COE followed by DVFE. Patients with tissue abnormalities found by COE or DVFE undergo biopsy within 2 weeks.
  Interventions: Procedure: fluorescence imaging; Procedure: biopsy; Procedure: examination
- Arm II - Comparison of surgical margins using COE vs. DVFE (Experimental): Comparison of surgical margins using COE vs. DVFE
  Interventions: Procedure: fluorescence imaging; Procedure: biopsy; Procedure: examination; Procedure: Comparison of surgical margins by COE vs. DVFE

INTERVENTIONS:
Procedure: fluorescence imaging — Undergo DVFE
Procedure: biopsy — Undergo scalpel biopsy
  Other Names: biopsies
Procedure: examination — Undergo COE
  Other Names: Exam; Medical Assessment; Medical Exam; Medical Examination; Medical Inspection
Procedure: Comparison of surgical margins by COE vs. DVFE — Surgical margin determination using DVFE
  Arms: Arm II - Comparison of surgical margins using COE vs. DVFE

SUMMARY:
This clinical trial studies direct visual fluorescence in finding oral cancer in high-risk patients and patients undergoing routine dental care. Diagnostic procedures, such as direct visual fluorescence, may help find and diagnose oral cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the diagnostic benefit of the VELscope (direct visual fluorescence) inspection in oral examination.

II. Efficacy of the VELscope in identifying dysplastic (premalignant) and malignant oral mucosal lesions and in discriminating these lesions from common benign tissue changes.

III. Accuracy of clinical judgment versus VELscope findings. IV. Ability of the VELscope to identify lesions or extent of lesions beyond what is clinically apparent.

OUTLINE:

Patients undergo conventional oral examination (COE) followed by direct visual fluorescence examination (DVFE). Patients with tissue abnormalities found by COE or DVFE undergo scalpel biopsy within 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIGH-RISK POPULATION:
* 33 consecutive consenting patients presenting to The Ohio State University James Cancer Hospital Otolaryngology Department with a suspicious oral lesion or prior biopsy-confirmed epithelial dysplasia (mild, moderate, severe), carcinoma in situ (CIS), or squamous cell carcinoma (SCC) will be recruited; adult patients presenting for initial evaluation for treatment planning and/or presenting for follow-up appointments monitoring for recurrence will be eligible to participate
* GENERAL POPULATION:
* 250 consecutive consenting patients presenting to The Ohio State University College of Dentistry for routing dental care will be recruited; adult patients presenting to the screening clinic for initial oral evaluation will be eligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-11-11 (Actual); Primary Completion 2016-10-03 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of DVFE compared to visual inspection by conventional oral examination alone | At the time of examination
  Will be evaluated by calculating sensitivity and specificity and their corresponding exact 95% confidence intervals. Association between the two techniques will be assessed using the simple kappa statistic.
Differences between lesional margins identified by COE and DVFE | At the time of examination
  Will be evaluated using the dependent t-test. In the event that the parametric requirements of this test are not met, the Wilcoxon, matched-pairs, signed-ranks test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin McNamara, DDS, MS, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu